CLINICAL TRIAL: NCT03480399
Title: Long Term Morbidity and Quality of Life After Multivisceral Resection for Primary Retroperitoneal Soft Tissue Sarcomas: a Prospective Observational Study
Brief Title: Long Term Morbidity and Quality of Life in Retroperitoneal Sarcomas
Acronym: LTM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Marco Fiore, Attending Surgeon, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Other Study IDs: INT13-14
Record Dates: First submitted 2016-09-07; First posted 2018-03-29 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Sarcoma, Soft Tissue; Retroperitoneal Neoplasms; Surgery; Quality of Life; Morbidity
Keywords: retroperitoneal sarcoma; quality of life; morbidity; surgery
MeSH Terms: conditions — Sarcoma; Retroperitoneal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
No prospective data exist about long term morbidity and quality of life after multivisceral surgical resection for retroperitoneal soft tissue sarcoma (RSTS).

In order to assess the safety of this surgical approach and the effect on the Quality of Life over the long period we propose a prospective observational study.

The hypothesis is that the surgical treatment has no significant impact in determining a lower Quality of Life in the long term.

Objectives Primary objective Estimate the difference between baseline and 4 and 12 months scores of the "global health status / QoL" scale in patients primarily treated for localized RSTS, as determined in QLQ-C30 version 3.0.

Secondary objectives

* Evaluate the long term morbidity of aggressive surgical approach to RSTS in terms of renal failure.
* Evaluate the difference between baseline and 4 and 12 months scores of DN4 / LEFS / BPI questionnaires.
* Evaluate the difference between baseline and 4 and 12 months scores of the following scales from QLC-C30: PF2, RF2, EF, CF, SF, FA, FI.
* Evaluate the difference between baseline and 4 and 12 months scores of the following scales and single items from QLC-C29: Blood and mucus in stool, Stool frequency, Sexual interest, Impotence, Dyspareunia.
* To correlate the surgical resection pattern (number and type of organs resected) and the tumor features (size, grading and histological subtype) with the long-term morbidity and quality of life.

Eligibility Inclusion criteria

* Adult patients (age > 18 years) with primary localized RSTS surgically treated at our institution
* Written, voluntary, informed consent

Exclusion criteria

- Recurrent disease

DETAILED DESCRIPTION:
Study description This is an observational study aimed to prospectively evaluate the long term morbidity of aggressive surgical approach to RSTS and the impact over the patients' quality of life. Consecutive patients candidate to surgery for primary RSTS will be offered to be enrolled. We plan to include all the RSTS patients consecutively operated on for primary retroperitoneal sarcoma from first accrual on up to the 24 months after the study start.

At the entrance of the study, an informed written consent will be obtained. Study participants will be asked to complete four self-filled in one-off questionnaires (see "Study parameters" paragraph).

Study parameters Study parameters EORTC QLQ-CR29 and EORTC QLQ C30 questionnaires (baseline, 4 mos, 12 mos) LEFS questionnaire (baseline, 4 mos, 12 mos) BPI questionnaire (baseline, 4 mos, 12 mos) DN4 questionnaire (baseline, 4 mos, 12 mos) Serum creatinin (baseline, 4 mos, 12 mos) Morbidity events (4 mos, 12 mos) Neurologic exam of lower limbs (baseline, 4 mos, 12 mos) Disease status (4 mos, 12 mos)

* In case of preoperatory complementary treatment, the questionnaires will be administrated just before the beginning of the treatment.

* Quality of Life: the core questionnaire, the EORTC QLQC30,is an extensively validated questionnaire for the assessment of health related quality of life in cancer patients (Aaronson 1991). It contains both functional (physical, role, cognitive, emotional, social), and physical symptom multidimensional scales (fatigue, pain, and nausea and vomiting) as well as two single item "global health status" and "quality of life" scales, plus several single-item symptom measures. The QLQ-CR29 is a condition specific module (colo-rectal disease) developed to be used in conjunction with EORTC QLQC30; it is made up of 29 items for a total of four scales assessing urinary frequency, faecal seepage, stool consistency and body image as well a number single items scales. Both the tools are available and validated in the Italian language.
* Femoral Impairment: the dedicated questionnaire (Lower Extremity Functional Scale - Italian Version, LEFS questionnaire) will investigated daily life activities that require ad adequate function of knee joint stability and quadriceps strength as a surrogate of motor impairment of homolateral femoral nerve.
* Chronic Pain Syndrome: the Italian version of the 'Brief Pain Inventory Short form" (BPI, attached) ( ) will be administered in order to obtain information on pain status at censored time (basal, 4 and 12 months after surgery values).
* Neuropathic Pain: the Italian version of "Douleur Neuropathique en 4 Questions" (DN4, attached) will be administered in order to obtain information on neuropathic pain at censored time (basal, 4 and 12 months after surgery scores).
* Long term morbidity: morbidity events will specifically regard femoral nerve impairment at physical examination, abdominal complications, sexual life and physiological functions. Renal failure in particular will be investigated by renal function blood tests monitoring and glomerular filtration rate (GFR) calculated according to Cockroft-Gault and simplified MDRD (Modification of Diet in Renal Disease) methods. Serum creatinine value will also be registered. Renal failure will be defined according to National Kidney Foundation 2002 criteria (Stage 2 or higher), and classified according to GFR thresholds.
* Disease status will be recorded and in case of local and/or distant relapse the date of events will also be retrieved.

Statistical considerations Statistical analyses

1. Primary end-point The two-sided 95% confidence interval (95%CI) of the paired difference between baseline and 4 (or12) months scores will be calculated for the primary outcome scale variables (items "29" and "30" QLQ-C30).
2. Secondary end-points Descriptive statistics and frequency tabulation were used to summarize patient characteristics and long term morbidity profile. Continuous variables will be described with appropriate summary statistics such as the mean, median, standard deviation, minimum and maximum. Categorical variables will be tabulated with frequencies and percentages. The probabilities of renal failure and femoral neuropathy will be estimated by the corresponding relative frequencies; their corresponding 95% confidence limits will be calculated using the exact method, i.e. taking into account the binomial distribution of proportions. The binary associations between the surgical resection pattern (number and type of organs resected) and the tumor features (size, grading and histological subtype) will be tested by using exact chi-square test. As regards the quantitative parameters measured over time, summary statistics (mean, median, standard deviation, minimum and maximum) or frequencies and percentages - as appropriate for the type of data - will be summarized by each time point; mixed models will be used to analyze the longitudinal measurements, allowing to take into account the within subject correlation and to straightforwardly analyze unbalanced data that may arise in the study.

Interim Analysis We plan to performed an interim cross-sectional analysis at the end of patient enrollment in order to describe the study population at baseline, according to the primary and secondary endpoints.

Sample size

We plan to include all the RSTS patients consecutively operated on for primary retroperitoneal sarcoma from first accrual on for the next 24 months (about 60 patients estimated.

A sample size of 60 patients allows the estimation of a two-sided 95,0% confidence interval for the paired difference between baseline and post treatment scores with a precision (half CI width) of 0.25 times the standard deviation of the difference.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients affected by primary retroperitoneal sarcoma and candidated to complete surgery (multivisceral resection)

Exclusion Criteria:

* Recurrent Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary retroperitoneal sarcoma candidated to multivisceral resection
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Global Health Status | 4 and 12 months postoperatively
  Change between baseline and 4 and 12 months scores of the "global health status / QoL" scale in patients primarily treated for localized RSTS, as determined in QLQ-C30 version 3.0.

SECONDARY OUTCOMES:
Renal failure | 12 months postoperatively
  Evaluate the long term morbidity of aggressive surgical approach to RSTS in terms of renal failure.
DN4 questionnaire for neuropathic pain | 4 and 12 months postoperatively
  Change between baseline and 4 and 12 months scores
LEFS questionnaire for lower limb function | 4 and 12 months postoperatively
  Change between baseline and 4 and 12 months scores
BPI questionnaire for chronic pain | 4 and 12 months postoperatively
  Change between baseline and 4 and 12 months scores
QLC-C30, Functional Scales | 4 and 12 months postoperatively
  Change between baseline and 4 and 12 months scores
QLC-C29 | 4 and 12 months postoperatively
  Change between baseline and 4 and 12 months scores

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fiore M, Brunelli C, Miceli R, Manara M, Lenna S, Rampello NN, Callegaro D, Colombo C, Radaelli S, Pasquali S, Caraceni AT, Gronchi A. A Prospective Observational Study of Multivisceral Resection for Retroperitoneal Sarcoma: Clinical and Patient-Reported Outcomes 1 Year After Surgery. Ann Surg Oncol. 2021 Jul;28(7):3904-3916. doi: 10.1245/s10434-020-09307-7. Epub 2020 Nov 11. PMID 33175262